CLINICAL TRIAL: NCT03126253
Title: The Burden of Childhood Anemia in Bangladesh:
Brief Title: The Burden of Childhood Anemia in Bangladesh: Does Socioeconomic Status Matter?
Status: Completed | Type: Observational
Sponsor: Shahjalal University of Science and Technology (Other)
Responsible Party: Principal Investigator, G.M. Rabiul Islam, Associate Professor, Shahjalal University of Science and Technology
Other Study IDs: FET-CA
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Anemia
Keywords: childhood anemia, socioeconomic status
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anemia — Hemoglobin level will be used as the parameter for diagnosing anemia. The HemoCue system was used to estimate the concentration of hemoglobin in capillary blood. WHO guidelines for the diagnosis of anemia that were adopted by the Demographic Health Surveys will be used in this study. Briefly, a hemoglobin concentration of less than 70 g/L will be consider to define severe anemia, 70-99 g/L for moderate anemia, and 100-109 g/L will be presumed to correspond to mild anemia. The above-mentioned classification of anemia as "severe" "moderate" and "mild" categories is based on blood hemoglobin cutoffs (will be adjusted for altitude and smoking) recommended by the Center for Disease Prevention of United States; this classification has also been adopted by the World Health Organization.

SUMMARY:
Childhood anemia is a global public health problem that is associated with life-threatening consequences such as growth retardation, impaired motor and cognitive development, and increased morbidity and mortality. Anemia can be caused by a variety of factors such as nutritional deficiencies (i.e., iron, folic acid, vitamin B12, and vitamin A), infections (i.e., helminth), and blood disorders (i.e., hemoglobinopathies). The World Health Organization (WHO) estimates that approximately 50% of anemia cases can be attributed to iron deficiency. This is an estimated global average that varies widely depending upon the location in question. The World Bank estimates for 2011 claim that approximately 55.60% of all Bangladeshi children under five years of age are suffering from anemia. The relationship between socioeconomic status (SES) inequality and anemia among the children has never been conclusively and it is unclear if the children of the age group of 6-59 months have uniformly high levels of anemia during all the stages of development, e.g., during the infant, toddler, and preschool stages. In addition, there is a dearth of evidence from Bangladesh, where the meaning of sociodemographic characteristics may be different from that in other countries. Therefore, this study attempts to fill the above-mentioned lacuna by investigating and evaluating the association of SES inequality, among other explanatory variables, on the development of childhood anemia during different stages of child development and to answer the questions: (a) Is SES a factor impeding childhood anemia along with other explanatory variables? (b) In which stage of child development, the chance of disparaging with childhood anemia is highest? (c) Is there evidence of between child development stages differences in the strength and form of association disparities between having childhood anemia and SES? (c) What are the predictive margins for SES-associated anemia in the case of infants, toddlers, and preschool children? The results of this analysis will be reported for elucidating the potential effects of SES and the stages of child development that are usually neglected in the conventional scientific literature. Moreover, as anemia is one of the current key health issues in Bangladesh, it is also expected that the findings of this study would contribute significantly toward shaping the health policy strategy of the country.

DETAILED DESCRIPTION:
The data collected by the 2011 Bangladesh Demographic Health Survey (BDHS), conducted by the National Institute for Population Research and Training (Ministry of Health and Family Welfare, Bangladesh), will be used for the purpose of this study. in the BDHS 2011, A nationally representative household-based sample was created through a stratified, multistage cluster sampling strategy in which 600 primary sampling units were constructed (207 in urban areas and 393 in rural areas). The primary sampling units were derived from a sampling frame created for the 2001 Bangladeshi census from seven divisions of Bangladesh. Households were selected randomly from each primary sampling unit. The data pertaining to the socioeconomic and sociodemographic factors were collected using a structured open-ended interview. The questionnaire used for this purpose was modeled on the MEASURE DHS questionnaires. Prior to the use, these questionnaires were adapted for the use in Bangladesh through a series of meetings with a Technical Working Group (TWG) that comprised of representatives from the National Institute of Population Research and Training (NIPORT,) Mitra and Associates, the International Centre for Diarrheal Diseases and Control in Bangladesh (ICDDR, B), USAID/Bangladesh, and MEASURE DH. The questionnaires were drafted in English and then translated into Bangla which is the national language of Bangladesh. The translations were reviewed by the experts as well as by the volunteers and a pilot study was conducted to validate the same. Of the total of 17,964 selected households, face-to-face interviews were successfully completed for 17,141 corresponding to a household response rate of 98%. The subjects for the examination of anemia were 2320 children aged 6-59 months, were raised from every third household of the BDHS sample. After excluding subjects with missing data, a total of 2068 individuals were selected for this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infant: Less than or equal to 12 months old
* Toddler: between 13-36 months
* Preschool children: between 37-59 month

Exclusion Criteria:

* Child 0-5 months

Ages: 6 Months to 59 Months | Sex: All
Age Groups: Child
Study Population: children 6-59 month of age in Bangladesh
Sampling Method: Non-Probability Sample
Enrollment: 2320 (Actual)
Dates: Start 2011-05-11 (Actual); Primary Completion 2011-07-08 (Actual); Study Completion 2012-01-18 (Actual)

PRIMARY OUTCOMES:
Anemia | Baseline
  Blood hemoglobin level will be used as the parameter for diagnosing anemia.

CONTACTS AND LOCATIONS:
Overall Officials: GM MI Islam, PhD, Principal Investigator — Shahjalal University of Science and Technology
Locations (1):
- Data analysis, Sylhet, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Islam GMR. Association of Socioeconomic Status With Childhood Anemia Among Infant, Toddler, and Preschool Children in Bangladesh. Value Health Reg Issues. 2020 May;21:141-148. doi: 10.1016/j.vhri.2019.09.008. Epub 2019 Dec 5. PMID 31812112
- See also: Report of the survey — https://dhsprogram.com/pubs/pdf/fr265/fr265.pdf
- Available data/document: Report of the survey along with sampling plan — https://dhsprogram.com/pubs/pdf/fr265/fr265.pdf